CLINICAL TRIAL: NCT05902403
Title: Risk Factors for Prolonged Mechanical Ventilation in Elevated Mean Airway Pressure Based on a Remote Ventilation Monitoring Platform
Brief Title: Risk Factors for Prolonged Mechanical Ventilation in Elevated Mean Airway Pressure
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RemoteVentilateView
Record Dates: First submitted 2023-06-04; First posted 2023-06-15 (Actual); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Mechanical Ventilation Pressure High; Intensive Care Unit

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Elevated Initial Mean Airway Pressure: Patients recieving invasive mechanical ventilation with mean airway pressure no less than 10 centimeter of water within the first 24 hours on ICU admission.
  Interventions: Other: invasive mechanical ventilation

INTERVENTIONS:
Other: invasive mechanical ventilation — Invasive mechanical ventilation for patients admitted to the ICU

SUMMARY:
This multicentric prospective clinical practice study aims at evaluating risk factors associated with a prolonged mechanical ventilation and other outcomes such as barotrauma and ICU length of stay in patients with elevated initial mean airway pressure based on a remote ventilation monitoring system which records venlitor input and output data (including waveforms).

DETAILED DESCRIPTION:
Brief Background:

Evidence has accumulated that protective lung ventilation and the patient-ventilator interaction are related to the outcome of patients with lung injury. While most current studies focus on the static parameters and their association with outcomes, dynamic ventilation parameters may provide a more comprehensive assessment than static ones. Time-varying features of ventilator parameters should be paid more attention. Recently, we have developed a remote mechanical ventilation visualization network system (RemoteVentilateView) and, simultaneously, a related automatic recognition algorithm for different types of patient-ventilator asynchrony. This system enables ventilation data fully used. Our main focus is on patients who have an average airway pressure no less than 10 cmH2O upon admission to the ICU. This population has a higher ventilation intensity and may be more at risk of ventilator-induce lung injury than the average ICU patients. We aims to identify risks factors associated with a prolonged mechanical ventilation and other outcomes such as barotrauma in this specific population.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving invasive mechanical ventilation, an average mean airway pressure ≥10 cmH2O for 6 consecutive hours within the first 24 hours of ICU admission.

Exclusion Criteria:

* Currently receiving or expected to receive ECMO treatment within 24 hours;
* Glasgow Coma Scale (GCS) score less than 8 due to cardiac arrest, traumatic brain injury, or acute stroke;
* Requiring invasive mechanical ventilation due to neuromuscular diseases;
* Exceeding 24 hours from ICU admission to connection to the remote monitoring system.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study enrolls patients admitted to ICU needing intubation and mechanical ventilation with elevated initial mean airway pressure.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-06-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
liberation from MV at day 7 | 7 days
  liberation from MV was defined as no need for MV at least 24 consecutive hours.

SECONDARY OUTCOMES:
Duration of mechanical ventilation and 28 days ventilator free days | 28 days
  Ventilator-free days (VFDs) were defined as a time frame of 28 days from intubation. For intubated patients, in caseof reintubation within 28 days, VFDs were counted from the last successful extubation. The use of non-invasive ventilation (NIV) after extubation was not considered as a ventilation period. Finally, zero VFDs were assigned to 28-day non-survivors, regardless of their intubation status.
Barotrauma | 7 days
  We consider as barotrauma within 7 days any pneumothorax, pneumomediastinum, subcutaneous emphysema or pneumatocele > 2cm detected on image exams between inclusion and 7 days, except those judged to be clearly caused by invasive procedures.
28-day Mortality | 28 days

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Qilu Hospital of Shangdong University, Jinan, Shandong
  - Sichuan Provincial People's Hospital, Chengdu, Sichuan
  - Shanghai Tenth People's Hospital, Shanghai

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Su L, Lan Y, Chi Y, Cai F, Bai Z, Liu X, Huang X, Zhang S, Long Y. Establishment and Application of a Patient-Ventilator Asynchrony Remote Network Platform for ICU Mechanical Ventilation: A Retrospective Study. J Clin Med. 2023 Feb 16;12(4):1570. doi: 10.3390/jcm12041570. PMID 36836113
- [Background] Urner M, Juni P, Hansen B, Wettstein MS, Ferguson ND, Fan E. Time-varying intensity of mechanical ventilation and mortality in patients with acute respiratory failure: a registry-based, prospective cohort study. Lancet Respir Med. 2020 Sep;8(9):905-913. doi: 10.1016/S2213-2600(20)30325-8. Epub 2020 Jul 28. PMID 32735841
- [Background] Chi Y, Zhang Q, Yuan S, Zhao Z, Long Y, He H. Twenty-four-hour mechanical power variation rate is associated with mortality among critically ill patients with acute respiratory failure: a retrospective cohort study. BMC Pulm Med. 2021 Oct 25;21(1):331. doi: 10.1186/s12890-021-01691-4. PMID 34696739
- [Background] Long Y, Su L, Zhang Q, Zhou X, Wang H, Cui N, Chai W, Wang X, Rui X, Liu D. Elevated Mean Airway Pressure and Central Venous Pressure in the First Day of Mechanical Ventilation Indicated Poor Outcome. Crit Care Med. 2017 May;45(5):e485-e492. doi: 10.1097/CCM.0000000000002290. PMID 28244940
- [Background] Su L, Pan P, Liu D, Long Y. Mean airway pressure has the potential to become the core pressure indicator of mechanical ventilation: Raising to the front from behind the clinical scenes. J Intensive Med. 2021 May 28;1(2):96-98. doi: 10.1016/j.jointm.2021.04.002. eCollection 2021 Oct. PMID 36788801
- [Background] McConville JF, Kress JP. Weaning patients from the ventilator. N Engl J Med. 2012 Dec 6;367(23):2233-9. doi: 10.1056/NEJMra1203367. No abstract available. PMID 23215559